# PRF Membrane and Recovery After Periapical Surgery: A 3D Imaging Study

PRF Membrane and Recovery After Periapical Surgery: A 3D Imaging Study

**Study Unique Protocol ID:** 

3736-1/2022/EKU

**NCT Number:** Not available

## Aim

Comparisation of the swelling, the quality of life and the post operative pain after endodontic surgery with and without of the use of A-PRF+.

## Matherials and methods

Patient selection:

• 10-10 per each group

#### **Inclusion Criteria:**

- Adults aged 20-65 years, both male and female.
- Diagnosed with periapical disease, including periapical cysts or granulomas.
- Requiring periapical surgery as part of their treatment plan.
- Presenting a tooth needing endodontic surgery with periradicular lesions of strictly endodontic origin.
- Size of the bone crypt between 6 mm and 12 mm.
- Non-surgical retreatment considered unfeasible or previously failed.
- Apical root canal free from posts over a length of at least 6 mm.
- Adequate coronal restoration without coronal leakage.
- Willing and able to provide written informed consent.
- Capable of attending follow-up visits and participating in required assessments.
- Maxillary and mandibular teeth limited to the 2nd premolar to 2nd premolar regions.
- Without general medical contraindications for oral surgical procedures.

#### **Exclusion Criteria:**

- Patients with systemic conditions affecting healing, such as:
  - Uncontrolled diabetes mellitus.
  - Autoimmune disorders.
  - Chronic inflammatory diseases.
- Pregnant or breastfeeding individuals.
- Use of medications or therapies that may interfere with healing, including:
  - o Bisphosphonates.
  - o Immunosuppressants.
  - Radiotherapy.
  - Oncological therapies (e.g., chemotherapy, immunotherapy).
- Requires antibiotic prophylaxis or therapy.
- History of allergies or adverse reactions to blood-derived products.
- Neuropsychiatric disorders.
- Active infection or severe periodontal disease in the surgical area.
- Periodontal probing depths greater than 5 mm.

- Moderate to severe periodontal bone loss.
- Vertical root fractures.
- Perforation of the furcation area or root canal, except for the apical area.
- Smokers or individuals unwilling to refrain from smoking during the study period.
- Participation in another clinical trial within the last 30 days.
- Absolute or relative contraindications for surgery.

## **Surgical procedure**

- If it is required and feasible endodontic treatment or retreatment maximum 1 week before surgery
- One surgeon perform all operation
- Local anaesthesia 2% lidocaine and ephinephrine 3x2 ml lidocaine
- Trapezoid submarginal flap (Ochsenbein-Luebke flap)
- 15 C surgical blade
- Ball shaped 0,27 mm diameter bone burr, 1:1 straight handpiece
- 3 mm of apical portion is resected- in one piece perpendicular to the long axis placed in sterile saline
- 3 mm retrograde cavity- with diamond coated ultrasonic instruments
- Micorbiological sample
- MTA retrograde RCfilling
- Mobilisation of the flap
- In the test group the resection cavity was filld and covered with A-PRF+ membrane
- Tension free flap closure with 3-0 Silc suture

# PRF preparation

- In the test group before surgery 3 or 2 (depends on size of the cavity) 10ml glass tubes without additives
- 1300 rpm for 8 min centrifugation (Harmonycom)
- Using an A-PRF Duo centrifuge (Process for PRF, Nice, France)
- Placed in sterile container (PRF Box, Process for PRF, Nice, France)

# Postoperative instruction

- Diclofecan 50mg (Cataflam 50mg) 2x1 per day, for 3 days
- Rinses with 0,12% Chlorehexidine twice a day for 1 week
- No postoperatic antibiotics was described
- Suture removal after 7 days

# **Evaluation**

- 3D optical scans (Einstar, Shining 3D) were recorded over two time period, T0 (preoperative scan), T1 (day 3 postoperatively)
- VAS (Visula Analogue Scale) pain was graded on a score to 0-10, 0 no pain, 10 maximum intesity of pain, for 7 days
- Likert scale based questionary: ranging from 0 to 4, 0 non 4 very much, for 7 days daily starts ont he operation day
  - Postoperativ limitations in function: Mouth opening, Chewing, Speaking, Sleeping,
    Daily routine, Work

### **Statistical Analisys**

# **Statistical Analysis Plan**

# 1. Study Objectives

## • Primary Objective:

o To assess the impact of PRF membrane on postoperative swelling and its relationship with quality of life dimensions and pain.

## • Secondary Objectives:

- o To compare quality of life (QoL) dimensions and pain levels pre- and post-intervention between the PRF membrane group and the control group.
- To investigate correlations between swelling (volume) and postoperative QoL dimensions.

## 2. Study Design

• **Type**: Preliminary comparative study.

## • Groups:

- o **PRF Membrane Group** (10 participants): Underwent apicoectomy with PRF membrane application.
- Control Group (10 participants): Underwent apicoectomy without PRF membrane.

#### 3. Outcome Measures

## 1. Primary Outcomes:

- Postoperative swelling (volume): Measured using standardized evaluation methods.
- Quality of Life (QoL) dimensions: Assessed using a questionnaire with subdimensions (e.g., physical function, pain impact, anxiety, sleep disturbance).

## 2. Secondary Outcomes:

- o Pain intensity: Measured using the Visual Analog Scale (VAS).
- o Correlations between swelling and QoL dimensions.

## 4. Statistical Methods

## 1. Descriptive Statistics:

- Mean ± standard deviation for continuous variables (e.g., QoL scores, pain, swelling volume).
- o Frequency and percentage for categorical variables.

# 2. Normality Testing:

• **Shapiro-Wilk test**: Conducted for each variable to determine whether parametric or non-parametric tests will be used.

## 3. Comparative Analyses:

# o Between Groups:

- Independent samples t-test for normally distributed data.
- Mann-Whitney U test for non-normally distributed data.

## Within Groups:

- Paired t-test for normally distributed pre- and post-intervention comparisons.
- Wilcoxon signed-rank test for non-normally distributed data.

## 4. Correlations:

 Spearman's or Pearson's correlation will be used to evaluate the relationship between swelling (volume) and QoL dimensions depending on data distribution.

## 5. Significance Threshold:

• A two-tailed **p-value** < **0.05** will be considered statistically significant.

# 5. Missing Data

- Missing data will be handled by:
  - Listwise deletion for analyses where missing data is minimal.
  - Sensitivity analysis if missing data exceeds 10%.

## 6. Software

• All statistical analyses will be performed using **SPSS** or **R** software.

# 7. Reporting

- Results will include:
  - o Comparative tables of pre- and post-intervention outcomes.
  - o Statistical significance levels for group comparisons.
  - o Correlation matrices for swelling and QoL dimensions.